CLINICAL TRIAL: NCT05288153
Title: Metformin Efficacy and Safety for Gastric Intestinal Metaplasia: a Randomized Controlled Trial
Brief Title: Metformin Efficacy and Safety for Gastric Intestinal Metaplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Clinical Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20212212-C-1
Record Dates: First submitted 2022-02-15; First posted 2022-03-21 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Gastric Intestinal Metaplasia
MeSH Terms: interventions — Metformin; Folic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the metformin group (Experimental): Patients in the metformin group shall receive oral metformin at 500 mg per day for 6 months.
  Interventions: Drug: Metformin
- the folate group (Active Comparator): Patients in the folate group shall receive oral folate at 5 mg three times a day for 6 months.
  Interventions: Drug: Folate

INTERVENTIONS:
Drug: Metformin — Subjects will be instructed to take one tablet(500mg) of metformin after breakfast every day, and to visit the hospital every 4 weeks for evaluation of the subjective symptoms and for receiving a new supply of medication.
  Other Names: Glucophage
  Arms: the metformin group
Drug: Folate — Subjects will be instructed to take one tablet(5mg) of folate three times every day, and to visit the hospital every 4 weeks for evaluation of the subjective symptoms and for receiving a new supply of medication.
  Arms: the folate group

SUMMARY:
Gastric intestinal metaplasia significantly increases the risk of gastric cancer. Metformin, a biguanide, which is widely used for treating diabetes mellitus, has recently been suggested to have a suppressive effect on tumorigenesis and cancer cell growth. The investigators devised a prospective randomized controlled trial to evaluate the chemopreventive effect of metformin against gastric intestinal metaplasia and the safety of this drug in non-diabetic gastric intestinal metaplasia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 18 to 75 years old;
2. Body mass index (BMI) ranged from 18.5 to 23.9 at enrollment;
3. IM patients with OLGIM stage Ⅱ-Ⅲ diagnosed by upper gastrointestinal endoscopy and histopathological biopsy within the last 3 months;
4. Patients without H. pylori infection confirmed by 13C-urea breath test (UBT) or patients with H. pylori infection who completed the bismuth-containing quadruple program and had confirmed successful eradication by 13C-UBT.

Exclusion Criteria:

1. History of diabetes mellitus (use of medication and/or HbA1c over 6.5%);
2. History of regular use (defined as at least once per week) of NSAIDs and/or aspirin;
3. History of stomach surgery (including endoscopic submucosal dissection and endoscopic mucosal resection) or previously diagnosed malignant tumor;
4. History of heart failure, renal failure, liver cirrhosis or chronic hepatic failure;
5. Patients with contraindications or allergies to the drugs in this study;
6. Breastfeeding or pregnancy;
7. History of substance abuse or alcohol abuse in the past 1 year;
8. Severe mental illness;
9. Refusal of drug treatment;
10. Refusal of signing informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of reversal and progression of gastric intestinal metaplasia | 6 months
  To evaluate the effects of the therapies, each subject was assigned a stage score before the therapy (A) and at the end point (B) according to OLGIM stages.

SECONDARY OUTCOMES:
Rate of reversal and progression of gastric atrophy | 6 months
  To evaluate the effects of the therapies, each subject was assigned a stage score before the therapy (A) and at the end point (B) according to OLGA stages.
Fasting blood glucose | 6 months
  Fasting blood glucose in mg/dL.
Fasting blood insulin | 6 months
  Fasting blood insulin in μU/mL.
HbA1c | 6 months
  HbA1c in a percentage form.
Total cholesterol | 6 months
  Total cholesterol in mg/dL.
LDL-cholesterol | 6 months
  LDL-cholesterol in mg/dL.
Blood urea nitrogen (BUN) | 6 months
  Blood urea nitrogen (BUN) in mg/dL.
Creatinine | 6 months
  Creatinine in mg/dL.
physical examination findings | 6 months
  Physical examination findings included weight in kilograms, height in meters and weight and height will be combined to report body mass index (BMI) in kg/m^2.

OTHER OUTCOMES:
Changes of gastric mucosal bile acid profile in metformin group before the therapy and at the end point. | 6 months
  Investigators evaluate the changes of gastric mucosal bile acid profile in metformin group before the therapy and at the end point according to the results of UPLC-MS/MS and pathological.
Changes of gastric microbiota in metformin group before the therapy and at the end point. | 6 months
  Investigators explore the changes of gastric microbiota in metformin group before the therapy and at the end point according to the results of 16s rRNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, PhD, Study Director — Xijing Hospital of Digestive Diseases
Locations (2):
- China (2):
  - Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li S, Li X, Zhu X, Zhao X, Qu X, Lin K, Yao N, Wang N, Chen M, Zhang L, Shi Y. Therapeutic effect of metformin on reversing gastric intestinal metaplasia. Chin Med J (Engl). 2025 Jun 16. doi: 10.1097/CM9.0000000000003675. Online ahead of print. PMID 40518567